CLINICAL TRIAL: NCT01470651
Title: Armodafinil for Patients Starting Hepatitis C Treatment
Brief Title: Armodafinil for Patients Starting Hepatitis C Virus Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: European Medicines Agency issued a drug/drug interaction: sofosbuvir/modafinil
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Judith G. Rabkin, PhD, Research Scientist VI, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/6285
Record Dates: First submitted 2011-10-13; First posted 2011-11-11 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-10

CONDITIONS: Hepatitis C
Keywords: HCV+; HCV treatment; Fatigue; patients starting alpha interferon/ribavirin treatment
MeSH Terms: conditions — Hepatitis C; Fatigue | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Armodafinil (Experimental): Active medication
  Interventions: Drug: Armodafinil
- Sugar pill (Placebo Comparator): Inactive pill, matched to look like active medication
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Armodafinil — 50mg - 250mg pills, taken each morning, for 14 weeks
  Other Names: Nuvigil
  Arms: Armodafinil
Drug: Sugar Pill — Inactive pill, matched to look like active medication
  Other Names: Placebo Comparator
  Arms: Sugar pill

SUMMARY:
Fatigue is one of the most common side effects of the treatment of hepatitis C infection with pegylated interferon and ribavirin, and is a major cause of treatment discontinuation. Armodafinil is an FDA approved stimulant medication for the treatment of narcolepsy and shift-work sleep disorder. This is a randomized placebo controlled study to determine whether patients assigned to armodafinil have fewer missed doses, dose reductions or treatment discontinuation due to side effects in the first 12 weeks of treatment for hepatitis C infection than do placebo patients. Placebo patients are offered 14 weeks of open label armodafinil after Week 12.

DETAILED DESCRIPTION:
Four million Americans have chronic hepatitis C (HCV), and 30% of HIV+ patients are co-infected with HCV. Until May 2011, the standard treatment for HCV was the combination of alpha interferon (injected weekly) and ribavirin (daily pills) (IFN/RBV) for 48 weeks in order to achieve sustained virologic remission (cure). HCV treatment initiation was low, often because of concern about severe treatment side effects as well as high rates of virologic failure. Among the minority of medically eligible HCV+ patients (with or without co-morbid HIV/AIDS) who actually began treatment with IFN/RBV, side effects cause substantial attrition (about 20% by Week 12, 40% by Week 24). The most common adverse events are flu-like symptoms, of which fatigue is most prominent. Depressed mood is also common (mostly somatic symptoms).

Two new medications, telaprevir and boceprevir (protease inhibitors) have been successful in treatment of HCV in clinical trials, and both were approved by the FDA for those patients with genotype 1 HCV, and are marketed as of May 2011. One of the new drugs will be added to the current regimen for genotype 1 infection. Because both drugs are protease inhibitors, which develop rapid resistance when administered alone, they must be added to the current standard of care rather than replace it. This is expected to vastly increase willingness of doctors to recommend treatment, and for patients to agree to treatment. The investigators expect that most hepatologists will recommend, and patients agree to the addition of one of these medications from now on. However, it should be noted that both commonly cause fatigue if it isn't already present because of HCV itself, or peginterferon or ribavirin. The major adverse event associated with telaprevir is rash, and with boceprevir, anemia.

This is a 14-week placebo controlled double blind trial of armodafinil for patients about to begin HCV treatment, starting armodafinil or placebo 2 weeks prior to initiation of HCV treatment. Patients are recruited from the hepatology clinics at the respective sites. Randomization is 1:1. Placebo patients who continue HCV treatment are offered 14 weeks of armodafinil starting at Week 12 of HCV treatment when the armodafinil/placebo blind is broken.

Patients will be seen weekly for the first 4 weeks to titrate armodafinil dose and manage side effects, if any, and then biweekly, with telephone contact on the intervening weeks through Week 12. After that, monthly telephone calls through Week 24 will be conducted with patients randomized to armodafinil, and biweekly visits with placebo patients beginning armodafinil at Week 12.

The primary outcome measures concern non-adherence to INF/RBV treatment: 1) missed doses; 2) dose reductions, and 3) attrition due to side effects. Secondary outcomes include ratings of fatigue on the Fatigue Severity Scale, depression on the Patient Health Questionnaire (PHQ-9), and quality of life on the Endicott Quality of Life Enjoyment and Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* HCV+ patients medically cleared for IFN/RBV treatment -HIV+ or HIV-
* Speaks English
* Able and willing to give informed consent
* Fecund women: use barrier method of contraception

Exclusion Criteria:

* Untreated and uncontrolled hypertension
* Left ventricular hypertrophy
* Currently taking stimulant medication
* Uncontrolled mental health problems including: MDD, suicidal or homicidal ideation, bipolar disorder, or schizophrenia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weiss, Ph.D., MS, Principal Investigator — Icahn School of Medicine at Mount Sinai; Stephen J. Ferrando, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Mount Sinai Medical Center, New York, New York
  - New York-Presbyterian/Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Inactive pill, matched to look like active medication
  Placebo Comparator: Inactive pill, matched to look like active medication
Period: Overall Study
Arm/Group | Armodafinil | Sugar Pill
Started | 13 | 13
Completed | 6 | 10
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Sugar Pill | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 53.77 [28 to 65] | 57.23 [36 to 70] | 55.5 [28 to 70]
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Medications Form
Description: The Medication Adherence Form was designed to assess any HCV medication dosing changes, including discontinuation, and the reasons for the changes. The form asks specifically about the HCV medications: pegylated interferon, ribavirin and Incivek (or Victrelis), as well as the study medication, armodafinil.
Time Frame: HCV medication adherence reported at 12 weeks
Population: Not all patients were given all medications, subjects are not factored in if they were not told to take a given drug.
Measure: Mean (Standard Error); unit: Percentage of doses missed
Arm/Group | Armodafinil | Sugar Pill
Number analyzed (Participants) | 6 | 10
Percentage of doses missed
  pegylated interferon | 0 (0) | 1.74 (1.16)
  ribavirin | 0 (0) | 3.24 (1.87)
  Incivek (or Victrelis): number analyzed (Participants) | 5 | 9
  Incivek (or Victrelis) | 4.95 (3.06) | 2.88 (1.14)
  Armodafinil or Placebo | 14.00 (9.34) | 8.02 (4.23)

2. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: Fatigue Severity Scale is a 9-item scale measures the impact of fatigue on everyday functioning (e.g. "fatigue interferes with my work, family or social life"). Response format is a 7-point Likert scale of agreement with a 1-week time frame. Total score is the sum of item scores and ranges from 9 to 63 points, with higher scores indicating greater fatigue. A score greater than 40 is considered to be a clinically significant level of fatigue. Scores on the scale correlate highly with other measures of fatigue, is sensitive to change, and is routinely used in studies of modafinil/armodafinil.
Time Frame: Biweekly for the first month, monthly thereafter
Measure: Mean (Standard Deviation); unit: FSS score (out of 63)
Arm/Group | Armodafinil | Sugar Pill
Number analyzed (Participants) | 6 | 10
FSS score (out of 63)
  Baseline | 23.29 (17.17) | 26.90 (15.34)
  Week 2 | 30.71 (16.16) | 36.60 (17.37)
  Week 4 | 37.14 (17.58) | 38.90 (15.26)
  Week 8 | 32.00 (20.93) | 40.00 (18.06)
  Week 12 | 31.71 (20.15) | 38.40 (16.290)

ADVERSE EVENTS:
Time Frame: Baseline readings were collected two weeks before randomization to placebo or Armodafinil until 16 weeks after randomization. Measurements weekly until post-randomization week 12 at which point they were taken every other week.
Description: Side effects form listed: Nervousness, Irritability, Headaches, Nausea, Insomnia, Shortness of Breath, Difficulty Concentrating, Appetite/weight loss, Taste change, Dry mouth, Diarrhea, muscle aches, rash, fever, rectal pain, and two "other" fields. Side effect onset was defined as a two point increase (on a 5 point scale) from baseline.
Arm/Group | Armodafinil | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 12/13 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Armodafinil (N=13) | Sugar Pill (N=13)
Nervousness (Psychiatric disorders) | 4/12 | 3
Insomnia (Psychiatric disorders) | 3/12 | 6
Shortness of Breath (Nervous system disorders) | 5 | 9
Appetite or weight change (Nervous system disorders) | 8 | 10
Taste Change (Nervous system disorders) | 5 | 10
Dry Mouth (Nervous system disorders) | 8 | 8
Diarrhea (Gastrointestinal disorders) | 5 | 6
Muscle Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Fever (Immune system disorders) | 5 | 10
Rectal Pain (Gastrointestinal disorders) | 3 | 8
Headaches (Nervous system disorders) | 9 | 10
Irritability (Psychiatric disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 7 | 7
Difficulty in Concentration (Psychiatric disorders) | 6 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 11
Dizzyness (Nervous system disorders) | 2 | 3
Tingling Feeling (Nervous system disorders) | 1 | 0
Lightheadedness (Vascular disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
feeling cold (Nervous system disorders) | 0 | 1
Sore Throat (General disorders) | 1 | 0
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1
Allergy Symptoms (Immune system disorders) | 0 | 1
Testicular Pain (Reproductive system and breast disorders) | 0 | 1
Emotional instability (Psychiatric disorders) | 0 | 1
Swollen Eyes (Eye disorders) | 1 | 0
Altered Sense of Smell (Gastrointestinal disorders) | 0 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
It is difficult to attribute side effects to Armodafinil or placebo given patients were undergoing Hepatitis C Treatment throughout the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No